CLINICAL TRIAL: NCT00339833
Title: The Effect of Salsalate Treatment on Insulin Sensitivity and Insulin Secretion in Obese Non-Diabetic Individuals
Brief Title: The Effects of Anti-Inflammatory Treatment on Insulin Resistance in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Clifton Bogardus, Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 999903121; 03-DK-N121 (Other: National Institutes of Health Clinical Center); 03-DK-N121 (Other: NIHCC)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-01

CONDITIONS: Type 2 Diabetes; Diabetes
Keywords: Salsalate; Insulin Resistance; Diabetes Mellitus; Inflammation; Diabetes; HCV
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance; Inflammation | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salsalate (Experimental): Salsalate (3g/day) for 7 days
  Interventions: Drug: Salsalate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salsalate — The intervention was salsalate (3g/day) for 7 days.
  Arms: Salsalate
Drug: Placebo — Identical placebo for 7 days.
  Arms: Placebo

SUMMARY:
This study, conducted at the Phoenix Indian Medical Center, Phoenix, Arizona, will determine whether reducing subclinical inflammation lessens insulin resistance in healthy, obese volunteers. The study findings may lead to new strategies for preventing type 2 diabetes. In diabetes, blood sugar is higher than normal and can result in serious medical problems, such as blindness and kidney failure. People with subclinical inflammation-inflammation that does not produce symptoms, such as fever, pain, or skin redness-are at increased risk for diabetes. Although the reasons for this are not completely understood, it is known that subclinical inflammation exacerbates insulin resistance, which is a cause of diabetes. Insulin is a hormone that helps control blood sugar, and when it does not work properly, the condition is known as insulin resistance.

Normal, healthy volunteers between 18 and 45 years old with a body mass index of at least 30 kg/m2 and who have subclinical inflammation (determined by blood tests) may be eligible for this study. Candidates must be non-smokers and must not have an alcohol or drug problem. Candidates will be screened with a medical history and physical examination, electrocardiogram, and blood and urine tests. Participants will maintain a standard diet and undergo tests and procedures during a 14-day inpatient stay at the Phoenix Indian Medical Center.

DETAILED DESCRIPTION:
In healthy subjects, low-grade inflammation, as measured by serum levels of cytokines or acute phase proteins, is positively associated with adiposity. Recent studies indicate that chronic low-grade inflammation in non-diabetic individuals may cause decline in insulin sensitivity and increases the risk of developing type 2 diabetes. It has been proposed that reduction of low-grade inflammation may reduce the risk of development of type 2 diabetes. In agreement with this hypothesis, the class of anti-inflammatory drugs called salicylates (such as aspirin) that influence a specific anti-inflammatory pathway have been found to decrease plasma glucose levels and increase insulin sensitivity in rodents as well as people with type 2 diabetes.

In the present study, we propose testing whether administration of the anti-inflammatory drug Salsalate improves insulin sensitivity in obese non-diabetic individuals and whether this improvement is related with a decrease in serum markers of inflammation. Subjects will be randomly assigned to two treatment groups: placebo or Salsalate (3g/d). An oral glucose tolerance test and a combined euglycemic/hyperglycemic clamp to assess insulin sensitivity and insulin secretion will be performed before and after seven days of treatment. Results of this study may help to identify novel strategies to prevent type 2 diabetes in high-risk groups.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age: Greater than 18 and less than 45 years.

Number: 44 completed studies (22 placebo, 22 Salsalate).

Sex: 22 Males and 22 Females.

BMI: Greater than or equal to 30 kg.m(2)

EXCLUSION CRITERIA:

* Age below 18 or above 45 years to minimize the risk of glucose clamp.
* Diabetes mellitus (as per 75 g OGTT, WHO 1999 criteria)
* Cardiovascular disease including: abnormal EKG, personal history of coronary heart disease;symptomatic angina pectoris or cardiac insufficiency as defined by NYHA; classification as functional class III or IV.
* Systolic blood pressure greater than 160mmHG and/or diastolic blood pressure greater than 100 mmHg and/or on antihypertensive therapy or resting heart rate greater than 90 bpm.
* Hematological disorder, including prolonged prothrombin time (normal range 10.9-12.9 sec) and partial thromboplastin time (24-36 sec) and thrombocytopenia (less than 150,000 mm(3)).
* Respiratory disease (including influenza, asthma)
* Allergies (including hay fever)
* Gastrointestinal (including peptic ulcer), hepatic or renal disease (ALT and AST greater than 3-fold above upper limit of normal range, creatinine greater than 1.3 mg/dl).
* Alcoholism, alcohol-induced autonomic neuropathy.
* Any endocrinological disorder, including hypopituitarism/pituitary dysfunctions or lesions, hypo/hyperthyroidism, insulinoma.
* CNS disease
* Psychosis or personal history of any psychiatric disorder.
* Taking medications within one month prior to beginning the study, including medications known to have pharmacological interactions with salicylates or that may affect insulin sensitivity and secretion (including salicylates, COX 1 and COX 2 inhibitors, warfarin, Beta-Blockers, phenothiazines, antidepressants, antiarrhythmic drugs, antimuscarinic drugs).
* Acute inflammation as assessed by history, physical and laboratory examination (subjects with C-reactive protein 2 standard deviations above the population mean will not be admitted). The population mean was calculated from subjects admitted at our research unit.
* Pregnant or lactating females or females on hormonal contraceptives.
* History of metabolic acidosis.
* Allergy to aspirin, other salicylates, or bleeding diathesis or currently on oral anticoagulants.
* Any current viral illness.
* Active cancer within 5 years prior to screening for the study.
* Positive urine drug screening test.
* Inability to provide informed consent.
* Smokers

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2003-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bogardus Clifton, MD, Principal Investigator — National Institues of Diabetes and Digestive and Kidney Disease
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Vozarova B, Weyer C, Hanson K, Tataranni PA, Bogardus C, Pratley RE. Circulating interleukin-6 in relation to adiposity, insulin action, and insulin secretion. Obes Res. 2001 Jul;9(7):414-7. doi: 10.1038/oby.2001.54. PMID 11445664
- [Background] Pratley RE, Wilson C, Bogardus C. Relation of the white blood cell count to obesity and insulin resistance: effect of race and gender. Obes Res. 1995 Nov;3(6):563-71. doi: 10.1002/j.1550-8528.1995.tb00191.x. PMID 8653533
- [Background] Pickup JC, Crook MA. Is type II diabetes mellitus a disease of the innate immune system? Diabetologia. 1998 Oct;41(10):1241-8. doi: 10.1007/s001250051058. PMID 9794114
- [Derived] Koska J, Ortega E, Bunt JC, Gasser A, Impson J, Hanson RL, Forbes J, de Courten B, Krakoff J. The effect of salsalate on insulin action and glucose tolerance in obese non-diabetic patients: results of a randomised double-blind placebo-controlled study. Diabetologia. 2009 Mar;52(3):385-93. doi: 10.1007/s00125-008-1239-x. Epub 2008 Dec 23. PMID 19104769

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment location: clinical research unit at the NIDKK (Phoenix, AZ, USA)
Pre-assignment Details: Upon admission, all participants were placed on a weight maintaining diet (containing 50% of energy as carbohydrate, 30% as fat and 20% as protein). Body composition was measured by dual-energy x-ray absorptiometry. At least 3 days after admission and after a 12 h overnight fast a 2-h 75 g OGTT was performed to exclude diabetes.
Groups:
- Placebo: Placebo for 7 days.
Period: Overall Study
Arm/Group | Salsalate | Placebo
Started | 28 | 26
Completed | 22 | 18
Not Completed | 6 | 8
Not completed — Withdrawal by Subject | 1 | 2
Not completed — toothache | 0 | 1
Not completed — indigestion | 0 | 1
Not completed — Chest pain | 0 | 1
Not completed — minor infection | 0 | 1
Not completed — Poor venous access | 2 | 2
Not completed — anaemia or excess drop in glycaemia | 2 | 0
Not completed — Error in data records | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Salsalate | Placebo | Total
Number analyzed (Participants) | 22 | 18 | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 29 (7) | 33 (8) | 31 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 10 | 9 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 0 | 1 | 1
  White | 3 | 3 | 6
  Native American | 19 | 14 | 33
Region of Enrollment [Number; unit: participants]
  United States | 22 | 18 | 40
BMI [Mean (Standard Deviation); unit: kg/m2] | 37 (5) | 38 (6) | 37.5 (5.5)
Body Fat [Mean (Standard Deviation); unit: % body fat] | 38 (6) | 38 (7) | 38 (6.5)
Fasting plasma glucose [Median (Standard Deviation); unit: mmol/l] | 5.11 (0.33) | 5.06 (0.33) | 5.09 (0.33)
2 hour plasma glucose [Mean (Standard Deviation); unit: mmol/l] | 6.67 (1.17) | 6.61 (1.83) | 6.64 (1.50)
Fasting plasma insulin [Median (Full Range); unit: pmol/l] | 80 [56 to 104] | 63 [49 to 90] | 76 [49 to 104]
Basal EGP [Mean (Standard Deviation); unit: micro-mol/(kg*min)] | 10 (2) | 11 (2) | 10.5 (2)
Clamp R_d [Median (Full Range); unit: micro-mol/(kg*min)] | 13 [11 to 15] | 16 [13 to 20] | 14 [11 to 20]

OUTCOME MEASURES:

1. Primary Outcome: Change in Fasting Plasma Glucose Concentration
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Salsalate | Placebo
Number analyzed (Participants) | 22 | 18
mmol/l | 4.7 (6.5) | 0.0 (3.7)

2. Primary Outcome: Change in the Average Serum Insulin Concentration During the Last 40 Min of Clamp
Time Frame: last 40 min of clamp
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | Salsalate | Placebo
Number analyzed (Participants) | 22 | 18
l/min | 0.15 (0.21) | -0.06 (0.23)

ADVERSE EVENTS:
Arm/Group | Salsalate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes